CLINICAL TRIAL: NCT02583022
Title: A Randomized, Open-label, Single Center, Investigator-initiated Clinical Study to Evaluate the Safety and Efficacy of PAC-14028 Cream in Subjects With Mild to Moderate Atopic Dermatitis
Brief Title: A Study to Evaluate the Safety and Efficacy of PAC-14028 Cream in Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRPV1-AD_IIT
Record Dates: First submitted 2015-09-30; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PAC-14028 cream 1.0% (Experimental): PAC-14028 cream 1.0%, Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 cream 1.0%
- PAC-14028 cream vehicle (Placebo Comparator): PAC-14028 cream vehicle, Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 cream vehicle
- Elidel cream 1% (Active Comparator): Elidel cream 1%, Twice daily for 4 weeks
  Interventions: Drug: Elidel cream 1%

INTERVENTIONS:
Drug: PAC-14028 cream 1.0% — Topical application
  Arms: PAC-14028 cream 1.0%
Drug: PAC-14028 cream vehicle — Topical application
  Arms: PAC-14028 cream vehicle
Drug: Elidel cream 1% — Topical application
  Arms: Elidel cream 1%

SUMMARY:
The study is a Phase II, single center, randomized, open-label, placebo-controlled study in male and female subjects, aged ≥ 20 years with mild to moderate atopic dermatitis. All subjects will receive BID topical applications of PAC-14028 cream or vehicle or Elidel cream for up to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 20 and 65 years old
* Patients with atopic dermatitis, diagnosed according to Hanifin and Rajka diagnostic criteria
* SCORAD (SCORing Atopic Dermatitis) Score less than 40

Exclusion Criteria:

* Patients presenting symptoms of systemic infection at screening
* Patients who had been treated with oral steroids, oral antibiotics, systemic phototherapy, or immunosuppressants within the last 1 month prior to the investigational product administration
* Patients who had been treated with topical steroids or antibiotics within the last 2 weeks prior to the investigational product administration
* Pregnant women or breastfeeding women
* Women of childbearing potential or women who are planning a pregnancy during the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
SCORing Atopic Dermatitis (SCORAD) index | Change from baseline at Day 28

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) score | Change from baseline at Day 7, 14 and 28
Success rate to pruritus treatment | Change from baseline at Day 7, 14 and 28
Eczema Area and Severity Index (EASI) score | Change from baseline at Day 7, 14 and 28
Each SCORAD index | Change from baseline at Day 7, 14 and 28
Transepidermal Water Loss (TEWL) level | Change from baseline at Day 7, 14 and 28
Skin Hydration level | Change from baseline at Day 7, 14 and 28
  Skin hydration was measured using the Corneometer

CONTACTS AND LOCATIONS:
Overall Officials: BeomJoon Kim, Professor, Principal Investigator — Department of Dermatology, Chungang University Hospital